CLINICAL TRIAL: NCT01954797
Title: Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe): Protocol of an Observational Study Accompanying a Randomized Controlled Trial
Brief Title: Biomarkers and Perfusion - Training-Induced Changes After Stroke
Acronym: BAPTISe
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Alexander H Nave, Dr, Charite University, Berlin, Germany
Other Study IDs: BAPTISe; BMBF-G.2.15 (Other Grant/Funding Number: G.2.15)
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Stroke
Keywords: Physical fitness; relaxation; stroke; cerebral ischemia; cerebral perfusion; biomarkers; MRI
MeSH Terms: conditions — Stroke; Brain Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will receive blood draws (whole blood) for blood biomarker analyses.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Physical Fitness: Patients from this group underwent 4 weeks of aerobic fitness training additional to normal supportive care, 5 times a week, for 50 minutes
- Relaxation: Patients of this group received 4-weeks of relaxation sessions additional to normal supportive care, 5 times a week, for 50 minutes.

SUMMARY:
The purpose of this observational study is to examine the effects of 4-weeks of physical fitness training in patients with subacute ischemic stroke on cerebral imaging and blood-derived biomarkers.

DETAILED DESCRIPTION:
This biomarker-driven study uses an observational design to examine a subgroup of patients in the randomized, controlled trial "Physical Fitness Training in Subacute Stroke" (PHYS-STROKE). In PHYS-STROKE, 215 patients with subacute stroke (hemorrhagic and ischemic) receive either 4-weeks of physical training (aerobic training, 5 times a week, for 50 minutes) or 4-weeks of relaxation sessions (5 times a week, for 50 minutes). A convenience sample of 100 of these patients with ischemic stroke will be included in BAPTISe and will receive magnetic resonance imaging (MRI) scans and blood tests before and after the PHYS-STROKE intervention. Imaging scans will address parameters of cerebral perfusion and vessel size imaging. Blood tests will determine several parameters such as immunity, inflammation (including neopterin, MMP-9), metabolism (including ApoCIII, oxidized LDL, HOMA-index, uric acid, CK-MB, cystatin c, and leptin), cytokines (osteopontin, adiponectin), and endothelial function (SDF1-alpha, ADMA, sICAM, sVCAM, E-selectin, P-selectin). Additionally, we will assess the association between functional outcomes (co-primary outcome measures of PHYS-STROKE) and biomarkers including imaging results.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years
* Diagnosis of subacute ischemic stroke (within 5-45 days after stroke onset)as determined by initial MRI/CT scan of the brain
* Cortical, sub-cortical, or brainstem affection
* Barthel Index (BI) <65 at inclusion
* Able to sit for at least 30 seconds (unsupported or supported, i.e., holding onto supports such as the edge of the bed)
* Ability to perform aerobic exercise, determined by by responsible physician
* Provision of written informed consent

Exclusion Criteria:

* Lacking ability to comply with study requirements
* Stroke due to intracranial haemorrhage
* Previous subarachnoid hemorrhage or other hemorrhagic stroke
* Progressive stroke
* Not able to receive magnetic resonance imaging scans, including perfusion imaging
* Unable to perform the required exercises due to medical, musculoskeletal, or neurological problems
* Required help of at least 1 person to walk before stroke due to neurological (e. g., advanced Parkinson's disease, Amyotrophic Lateral Sclerosis, Multiple Sclerosis) or non-neurological co-morbidities (e. g. heart failure, orthopaedic problems)
* Life expectancy < 1 year as determined by responsible physician
* Drug or alcohol addiction within the last six months
* Significant current psychiatric illness defined as medication-refractory of bipolar affective disorder, psychosis, schizophrenia or suicidality
* Current participation in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited for this study are collected at the rehabilitation hospital and are participating in the PHYS-STROKE trial.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Cerebral perfusion | baseline and 4-weeks
  Magnetic resonance imaging (MRI)-based cerebral perfusion are assessed before and after the 4-weeks of physical fitness training.
  Primary and secondary endpoints are specified after completion of the interim analysis after inclusion of the first 24 patients (first stage). In a second stage the study is conducted with specified primary and secondary endpoints with recruitment of up to 76 remaining patients.
Blood-derived biomarkers | baseline and 4-weeks
  Changes in blood biomarkers are assessed before and after the 4-weeks intervention of physical fitness training.
  Primary and secondary endpoints are specified after completion of the interim analysis after inclusion of the first 24 patients (first stage). In a second stage the study is conducted with specified primary and secondary endpoints with recruitment of up to 76 remaining patients.

SECONDARY OUTCOMES:
next cerebrovascular event | 6 months
  Patients re-admitting hospital with suspected transient ischemic attack (TIA), stroke, or other cerebrovascular event within 6 months post stroke
functional outcome | directly after the end of intervention and 3 months post stroke
  functional outcome assessed via functional scores such as Barthel Index and walking speed (co-primary endpoints of PHYS-STROKE) as well as the modified Rankin Scale (mRS)

OTHER OUTCOMES:
functional outcome | 3 months
  Analyzing how changes in imaging measures and blood-derived biomarkers are related to each other and to differences in functional outcome, in particular gait speed, Barthel index (co-primary endpoints of PHYS-STROKE) and modified Rankin Scale
endothelial function assessment | measurement before and after the 4 weeks intervention
  the endothelial function of included patients will be assessed prospectively before and after the 4 week intervention with the Endopat2000 device. First measurement was conducted in January 11th 2014. Results will be correlated with imaging and blood-derived biomarkers as well as differences between intervention groups.
Clinical biomarkers including vital Parameters | measurements at baseline and all follow-up time points (measurement before and after the 4 weeks intervention, at 3 months and at 6 months after stroke)
  systolic and diastolic blood pressure, resting heart rate, body-mass-index, and waist-to-hip-ratio over time compared between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Martin Ebinger, MD, Principal Investigator — Center for Stroke Research Berlin; Alexander H Nave, MD, Principal Investigator — Center for Stroke Research Berlin
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rios AS, Temuulen U, Khalil AA, Villringer K, Ali HF, Akdeniz A, Grittner U, Becher M, Rackoll T, Nave AH, Sperber PS, Liman TG, Otte C, Endres M, Kufner A. Lesion-Network Mapping of Poststroke Depressive Symptoms: Evidence From Two Prospective Ischemic Stroke Cohorts. Stroke. 2025 Sep;56(9):2527-2539. doi: 10.1161/STROKEAHA.125.051858. Epub 2025 Jul 7. PMID 40620229
- [Derived] Jodicke RA, Huo S, Krankel N, Piper SK, Ebinger M, Landmesser U, Floel A, Endres M, Nave AH. The Dynamic of Extracellular Vesicles in Patients With Subacute Stroke: Results of the "Biomarkers and Perfusion-Training-Induced Changes After Stroke" (BAPTISe) Study. Front Neurol. 2021 Nov 8;12:731013. doi: 10.3389/fneur.2021.731013. eCollection 2021. PMID 34819906
- [Derived] Muller S, Kufner A, Dell'Orco A, Rackoll T, Mekle R, Piper SK, Fiebach JB, Villringer K, Floel A, Endres M, Ebinger M, Nave AH. Evolution of Blood-Brain Barrier Permeability in Subacute Ischemic Stroke and Associations With Serum Biomarkers and Functional Outcome. Front Neurol. 2021 Oct 20;12:730923. doi: 10.3389/fneur.2021.730923. eCollection 2021. PMID 34744972
- [Derived] Nave AH, Krober JM, Brunecker P, Fiebach JB, List J, Grittner U, Endres M, Meisel A, Floel A, Ebinger M. Biomarkers and perfusion--training-induced changes after stroke (BAPTISe): protocol of an observational study accompanying a randomized controlled trial. BMC Neurol. 2013 Dec 11;13:197. doi: 10.1186/1471-2377-13-197. PMID 24330706

DOCUMENTS (1):
  • Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT01954797/SAP_000.pdf